CLINICAL TRIAL: NCT05108220
Title: A Retrospective Cohort Study to Evaluate the Effects of Cannabidiol (CBD)-Containing Test Products on Anxiety Among Women in the U.S.
Brief Title: Evaluation of Effects of CBD Products on Anxiety Among U.S. Women
Status: Completed | Type: Observational
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00054510
Record Dates: First submitted 2021-06-04; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Anxiety; Generalized Anxiety Disorder
Keywords: Cannabidiol; Tetrahydrocannabinol; Anxiety; Women
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Cannabidiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- R-101: CBD oil, 30 mg CBD per serving, 0% THC per serving, medium-chain triglyceride dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-102: CBD oil, 20 mg CBD per serving, 0% THC per serving, medium-chain triglyceride dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-103: CBD oil, 30 mg CBD per serving, <0.3% THC per serving, medium-chain triglyceride dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-104: CBD oil, 20 mg CBD per serving, <0.3% THC per serving, medium-chain triglyceride dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-105: CBD capsule, 15 mg CBD per serving, 0% THC per serving, Rice Powder and Piperine dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-106: CBD capsule, 25 mg CBD per serving, 0% THC per serving, Rice Powder and Piperine dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-107: CBD capsule, 15 mg CBD per serving, <0.3% THC per serving, Rice Powder and Piperine dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- R-108: CBD capsule, 25 mg CBD per serving, <0.3% THC per serving, Rice Powder and Piperine dilution, carbon dioxide extraction method
  Interventions: Dietary Supplement: Cannabidiol (CBD)- containing consumer products
- Control: Waitlist control; no product

INTERVENTIONS:
Dietary Supplement: Cannabidiol (CBD)- containing consumer products — Oils or capsules containing CBD which could be purchased commercially within the U.S.
  Groups: R-101; R-102; R-103; R-104; R-105; R-106; R-107; R-108

SUMMARY:
The investigators will conduct a retrospective cohort analysis of a consumer trial conducted by Rae Wellness. The trial took place between October 15, 2020 and December 30, 2020 and involved 1350 U.S. women who used in-home use tests (IHUT) of various Cannabidiol (CBD) products. Participants were randomized to one of 9 groups: 8 groups received one of 8 different CBD products in the mail, and one group served as the control and did not consume any CBD product. The CBD products varied by method of delivery, concentration of Tetrahydrocannabinol (THC), and dosage of CBD. Participants were asked to use the product once daily for 60 day and to complete health questionnaires at baseline, 30 days and 60 days.

DETAILED DESCRIPTION:
Between October 1-7, 2020, women from across the US were recruited by Rae Wellness to participate in a 60-day in-home use test (IHUT) of various Cannabidiol (CBD) products. The inclusion criteria were: women; between the ages of 24-44; reported symptoms associated with at least 4 out of 6 health issues (stress; anxiety; pain; sleep issues; digestive issues; low libido). Individuals were excluded if they were pregnant or breastfeeding. 1,350 women were randomly selected to participate in the study. The participants were randomized to one of 9 groups in the IHUT (150 in each group): 8 groups received one of 8 different CBD products in the mail, and one group served as the control and did not consume any CBD product. The CBD products varied by method of delivery (oil or capsule), concentration of Tetrahydrocannabinol (THC; less than 0.3% THC or 0% THC), and dosage of CBD (15, 20, 25 and 30 mg). Participants were asked to use the product once daily every day for 60 consecutive days, and to complete a health questionnaire online on 3 occasions: before initiating the product (baseline), 30 days after initiating the product, and 60 days after initiating the product. Those in the control group were also asked to complete the health questionnaire at each time point but did not receive nor consume any CBD product. The health questionnaire assessed anxiety, physical health, digestive health, sleep patterns, general wellness and sexual satisfaction using questions drawn from validated health indices.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified female
* Ages of 24 to 44 years
* Reported symptoms associated with at least 4 out of 6 health issues (stress; anxiety; pain; sleep issues; digestive issues; low libido).

Exclusion Criteria:

-Pregnant or breastfeeding

Ages: 24 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified as female at enrollment
Study Population: 1350 women from across the United States
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | 60 days
  Anxiety score, according to the Generalized Anxiety Disorder (GAD)-7 scale. Scores range from 0 to 21, with higher scores representing more severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Rae Wellness PBC, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No